CLINICAL TRIAL: NCT02423577
Title: A Phase 2a, Randomized, Double-blind, Placebo-controlled Assessment of the Safety and Protective Efficacy of FF-3 Dry Powder Administered by Nasal Inhalation for 5 Days to Healthy Adult Subjects Who Are Experimentally Infected With a Challenge Strain of Influenza A Virus
Brief Title: Safety and Protective Efficacy of FF-3 Dry Powder in Healthy Subjects Infected With Influenza Challenge Strain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Autoimmune Technologies, LLC (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AIT02-2001; 2015-001103-31 (EudraCT Number); HHSN272201400003C (Other Grant/Funding Number: National Institute of Health, NIAID); DMID 14-0052 (Other: Division of Microbiology and Infectious Diseases)
Record Dates: First submitted 2015-04-19; First posted 2015-04-22 (Estimated); Results first posted 2017-08-14 (Actual); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Influenza
Keywords: antiviral; influenza; challenge
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FF-3 dry powder (Experimental): FF-3
  Interventions: Drug: FF-3 dry powder
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FF-3 dry powder — FF-3 dry powder administered by nasal inhalation
  Arms: FF-3 dry powder
Drug: Placebo — Placebo dry powder administered by nasal inhalation
  Arms: Placebo

SUMMARY:
The purpose of this study are to determine the effect FF-3 in comparison to placebo in subjects who are experimentally inoculated with a live, challenge strain of influenza A virus.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and non-pregnant, non-lactating female subjects of 18 to 50 years of age inclusive
2. Body Mass Index (BMI) of 18 to 32 kg/m2 inclusive and body weight of 50 to 110 kg inclusive.
3. Normal spirometry values at Screening and Baseline
4. Post-menopausal women with amenorrhea for at least 2 years will be eligible
5. Females of childbearing potential must use two acceptable birth control methods throughout the study and for 30 days after the last dose of the IMP:
6. Male subjects:

   * Must agree to use a condom (or diaphragm) plus spermicide in female partner) from the time of the first dose of IMP through 90 days after the last dose.
   * Must agree to not donate sperm for 90 days after the last dose of IMP.
   * Documented evidence of vasectomies in males for 180 days minimum prior to the first dose of the IMP is an acceptable form of contraception.
   * Males who claim abstinence as their method of contraception are allowed provided they agree to use a double barrier method (diaphragm plus spermicide in female partner or condom) should they become sexually active from screening to 90 days after the last dose of IMP.
7. Willing and able to provide written informed consent.
8. Willing and able to adhere to the lifestyle guideline restrictions outlined in the protocol

Exclusion Criteria:

* Subjects may not be enrolled in the study if any of the following exclusion criteria are fulfilled:

  1. Evidence of or history of clinically significant oncologic, pulmonary, hepatic, gastrointestinal, cardiovascular, hematologic, metabolic, neurological, immunologic, nephrologic, endocrine , or psychiatric disease.
  2. Current infection of any nature unless agreed as insignificant to the study by the Investigator and Medical Monitor.
  3. Nasal abnormalities, including nasal septum deviation, septum perforations, or polyps; history of recurrent epistaxis; history of sinus surgery and/or persistent hypertrophic inferior turbinates.
  4. Significant abnormalities at screening in safety laboratory tests, ECGs, or spirometry.
  5. Broncho-reactive airway disease (asthma, chronic obstructive pulmonary disease, current allergic rhinitis, cystic fibrosis, chronic bronchitis, emphysema). Individuals with a history of childhood asthma are not necessarily excluded and acceptable for screening.
  6. History of significant nasal irritation from use of nasal sprays or drops.
  7. History of drug or alcohol abuse within the past 2 years
  8. Nicotine product users
  9. Received an investigational drug or participated in another research study within 90 days of the first dose of IMP.
  10. Participated in a previous investigational study of FF-3.
  11. History of influenza vaccination with a live or attenuated vaccine within the previous year
  12. Use of prescription drugs within 14 days prior to the first dose of IMP, excepting oral contraceptives.
  13. Received any non-prescription medications, vitamins, or dietary supplements within 14 days of administration of the first dose of IMP, unless both the Principal Investigator and the Medical Monitor grant prior approval. Herbal supplements must be discontinued 7 days prior to the first dose of IMP.

  15. Tested positive for alcohol at screening or admission to the CRU. 16. Positive urine pregnancy test at the Screening Visit or positive serum pregnancy test on admission to the CRU (females only).

  17. Positive test for HIV, hepatitis B surface antigen (HBsAg) or anti-hepatitis C virus (anti-HCV) at the screening visit.

  18. Positive urine drug test at the screening visit or at admission to the CRU. 19. Likelihood of requiring treatment during the study period with drugs not permitted by the study protocol.

  20. Subjects who have donated blood or experienced other significant blood loss within 56 days of screening for the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 79 (Actual)
Dates: Start 2015-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Quintiles Drug Research Unit, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Potential subjects were screened to determine their susceptibility to infection with the challenge strain as indicated by a serum antibody titre less than 1:10. Only subjects susceptible to the challenge strain qualified for study specific screening.
Period: Overall Study
Arm/Group | FF-3 Dry Powder | Placebo
Started | 53 | 26
Completed | 53 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FF-3 Dry Powder | Placebo | Total
Number analyzed (Participants) | 53 | 26 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 53 | 26 | 79
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 25
  Male | 40 | 14 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 49 | 23 | 72
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 3 | 0 | 3
  White | 43 | 22 | 65
  More than one race | 5 | 2 | 7
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 53 | 26 | 79

OUTCOME MEASURES:

1. Primary Outcome: Frequencies of Viral Shedding
Description: Percentage of Subjects Demonstrating Viral Shedding.
Time Frame: Day 2 to Day 10
Population: The percentage of subjects demonstrating viral shedding was estimated for each treatment with corresponding asymptotic 95% confidence intervals, based on the normal approximation to the binomial distribution (Wilsons's method)
Measure: Count of Participants; unit: Participants
Arm/Group | FF-3 Dry Powder | Placebo
Number analyzed (Participants) | 53 | 26
Participants | 51 | 22
Statistical Analysis 1: Comparison: FF-3 Dry Powder vs Placebo; Test type: Superiority; p = 0.1436, Chi-squared; Risk Ratio (RR) = 1.14, 90% CI 2-sided [0.98 to 1.31]

ADVERSE EVENTS:
Arm/Group | FF-3 Dry Powder | Placebo
All-Cause Mortality (participants affected / at risk) | 0/53 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/26
Other Adverse Events (participants affected / at risk) | 46/53 | 23/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FF-3 Dry Powder (N=53) | Placebo (N=26)
Limb injury (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (6)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 7 (8)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Lethargy (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 5 (5) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1) | 2 (2)
Restless Legs Syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 1 (1) | 0 (0)
Influenza Like Illness (General disorders) | 34 (36) | 14 (14)
Vessel Puncture Site Haematoma (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1)
Medical device site rash (General disorders) | 0 (0) | 1 (1)
Feeling Hot (General disorders) | 0 (0) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (General disorders) | 2 (2) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Paraesthesia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Otitis Media (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes